CLINICAL TRIAL: NCT05330611
Title: Treatment of Adult Traumatic Rib Fractures With Percutaneous Cryoneurolysis for Pain Control (Trauma-PC2-study)
Brief Title: Treatment of Adult Traumatic Rib Fractures With Percutaneous Cryoneurolysis
Acronym: Trauma-PC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Joseph Forrester, Assistant Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64713
Record Dates: First submitted 2022-03-11; First posted 2022-04-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-08

CONDITIONS: Rib Fractures
Keywords: Percutaneous Cryoneurolysis
MeSH Terms: conditions — Rib Fractures | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The investigators are proposing a prospective, randomized trial evaluating efficacy of ultrasound-guided cryoneurolysis for pain control after traumatic rib fractures in patients 18-64 years of age.
  Eligible patients would be enrolled by the trauma service after consent is obtained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ultrasound-guided Cryoneurolysis: Group A (Experimental): Patients who are admitted to the Emergency Department after a traumatic injury. Patients will have rib fractures in any of ribs 3-9. Patients will be 18-64 years of age and will be randomized (1:1) to the ultrasound-guided cryoneurolysis group within 72 hours of admission to the ED.
  Intervention is ultrasound-guided cryoneurolysis of intercostal nerves creating lost lasting pain relief. Device used for cryoneurolysis is Iovera Smart tip 190
  Interventions: Device: Cryoneurolysis of Intercostal Nerves
- Standard-of-Care : Group B (Active Comparator): Patients who are admitted to the Emergency Department after a traumatic injury. Patients will have rib fractures in any of ribs 3-9. Patients will be 18-64 years of age and will be randomized (1:1) to Standard of Care which typically includes multi-modal pain therapy and pulmonary toilet.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Cryoneurolysis of Intercostal Nerves — Patients will be offered a minimally invasive intervention procedure for pain control called cryoneurolysis using an ultrasound-guided device called the Iovera Smart Tip 190.
  The direct application of cold to the intercostal nerves via Iovera device produces lesions in peripheral nervous tissue to block the pain caused by rib fractures.
  This procedure is particularly beneficial for patients who are not candidates for surgical stabilization of their rib fractures.
  Application of cryoneurolysis as an analgesic will reduce the amount of narcotics patients might need and instead provide them short- or long-term pain control with minimal risk.
  Follow up includes pain surveys administered in Chest Wall clinic or via telephone at 30, 90, 365 days post discharge.
  Arms: Ultrasound-guided Cryoneurolysis: Group A
Other: Standard of Care — Patients will be provided regular standard of care at the Stanford Hospital with short- or long-term follow-up provided at the Stanford Center for Reconstruction after Chest Wall Injury.
  Standard of care for patients with rib fractures that are not eligible for surgical stabilization includes multi-modal pain therapy and pulmonary toilet.
  Follow up includes pain surveys administered in Chest Wall clinic or via telephone at 30, 90, 365 days post discharge.
  Arms: Standard-of-Care : Group B

SUMMARY:
The purpose of this research study is to examine the effectiveness of using the Iovera Smart Time 190, for ultrasound-guided cryoneurolysis, in trauma patients 18-64 years old with rib fractures that are not candidates for surgical stabilization. This will offer patients the benefits of cryoneurolysis of the intercostal nerves, thereby providing short and long term pain control while their ribs heal.

The Iovera Smart Tip 190 is FDA approved for cryoneurolysis.

DETAILED DESCRIPTION:
The purpose of this research study is to examine the effectiveness of using the Iovera Smart Time 190, for minimally invasive ultrasound-guided cryoneurolysis, in trauma patients 18-64 years old with rib fractures that are not candidates for surgical stabilization. This procedure will offer patients the benefits of cryoneurolysis (freezing) of the intercostal nerves, thereby providing short and long term pain control while their ribs heal.

Patients in the intervention arm will receive cryoneurolysis via the Iovera device and patients in the control arm will receive standard of care which typically includes multimodal pain therapy and pulmonary toilet. Short and long term pain relief will be compared among both arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 64 years with any acute rib fracture between rib 3 and rib 9
* Pain score equal to or greater than 5 with deep inspiration
* Presenting and admitted to Stanford Adult Emergency Department, having a trauma consult, and being admitted to the trauma floors of Stanford Healthcare (SHC) for their inpatient stay

Exclusion Criteria:

* Radiographic evidence of metastasis to ribs
* Glasgow Coma Scale (GCS) score <13
* Patients undergoing SSRF (Surgical stabilization of rib fractures)
* Rib fractures located < 3cm from spinous process
* Coagulopathy (INR >1.5, Plt < 100)
* Other factors precluding cryoneurolysis at the attending's discretion
* If only ribs broken are 1,2 or 10,11,12
* Inability to be positioned for the procedure
* If the patient has the following conditions that the manufacturer of the Iovera device advises AGAINST using the device if present: Cryoglobulinemia, Paroxysmal cold hemoglobinuria, Cold urticaria, Raynaud's disease, open and/or infected wounds at or near the treatment site.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Daily Numeric Pain Score | At time of discharge from hospital (up to 1 month)
  Patients will be asked to verbalize their numeric pain score, measured on a scale of 0 to 10, with 0 being no pain and 10 being the worst pain.
  Daily numeric pain score is collected on the Day the patient is discharged from the hospital.

SECONDARY OUTCOMES:
Daily Narcotic Equivalents | Collected at discharge (up to 1 month), 1, 3, 12 months post discharge
  Morphine Milligram Equivalents (MME)
30-day mortality | Evaluated 1 month after hospital discharge
  Will be obtained from chart review after discharge
Need for ICU admission | 1 month after hospital discharge
  Will be obtained from chart review after discharge
30-day rib-specific admission | 1 month after hospital discharge
  Incidence of rib-specific readmission (delayed hemothorax, pneumothorax, pneumonia, pain)
The McGill Pain Questionnaire (MPQ) and Pain Rating Index (PRI) Scale Score | Collected 1, 3, 12 months (post hospital discharge)
  The McGill Pain Questionnaire (MPQ) is a validated 20 question instrument to quantify subjective pain and the scoring system yields a Pain Rating Index (PRI) score between Mild, Moderate or Severe. The questionnaire will be administered to the patient by study/clinical staff during follow up. The scoring system yields a pain rating index (PRI) score between 0 and 50 used to temporally track pain, higher scores correspond to higher pain levels.
The Glasgow Outcome Scale Extended (GOS-E) Score | Collected 1, 3, 12 months post hospital discharge
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery. The Extended GOS (GOSE) provides more detailed categorization into eight categories by subdividing the categories of severe disability, moderate disability and good recovery into a lower and upper category:
  1. Death (D)
  2. Vegetative state (VS)
  3. Lower severe disability (SD -)
  4. Upper severe disability (SD +)
  5. Lower moderate disability ( MD -)
  6. Upper moderate disability ( MD +)
  7. Lower good recovery (GR -)
  8. Upper good recovery (GR +)
  The questionnaire will be administered to the patient by study/clinical staff during follow up.
Short Form (SF-12) Health Survey Scale Score | Collected 1, 3, 12 months (post hospital discharge)
  The 12-Item Short-Form Health Survey is a widely used composite score used to gauge overall health. The composite score is based on 8 domains scores contained in the SF-12 questionnaire, which will be administered to the patient by study/clinical staff during follow up.
  Score ranges from 1 (Excellent) to 5 (Poor) , 1 (Yes, limited a lot) to 3 (No, not limited at all), 1 (Yes) 2 (No), 1 (Not at all) to 5 (Extremely), 1 (All of the time) to 6 (None of the time) and 1 (All of the time) to 5 (None of the time).
Length of hospital stay | Up to 1 month from ED arrival
  The length of hospital stay will be obtained from the patient's chart after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Forrester, MD, Principal Investigator — Stanford University; Ariel Knight, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Sharma OP, Oswanski MF, Jolly S, Lauer SK, Dressel R, Stombaugh HA. Perils of rib fractures. Am Surg. 2008 Apr;74(4):310-4. doi: 10.1177/000313480807400406. PMID 18453294
- [Background] Marasco S, Lee G, Summerhayes R, Fitzgerald M, Bailey M. Quality of life after major trauma with multiple rib fractures. Injury. 2015 Jan;46(1):61-5. doi: 10.1016/j.injury.2014.06.014. Epub 2014 Jun 21. PMID 25069400
- [Background] Fabricant L, Ham B, Mullins R, Mayberry J. Prolonged pain and disability are common after rib fractures. Am J Surg. 2013 May;205(5):511-5; discusssion 515-6. doi: 10.1016/j.amjsurg.2012.12.007. PMID 23592156
- [Background] Gordy S, Fabricant L, Ham B, Mullins R, Mayberry J. The contribution of rib fractures to chronic pain and disability. Am J Surg. 2014 May;207(5):659-62; discussion 662-3. doi: 10.1016/j.amjsurg.2013.12.012. Epub 2014 Jan 31. PMID 24612969
- [Background] Liman ST, Kuzucu A, Tastepe AI, Ulasan GN, Topcu S. Chest injury due to blunt trauma. Eur J Cardiothorac Surg. 2003 Mar;23(3):374-8. doi: 10.1016/s1010-7940(02)00813-8. PMID 12614809
- [Background] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Background] Todd SR, McNally MM, Holcomb JB, Kozar RA, Kao LS, Gonzalez EA, Cocanour CS, Vercruysse GA, Lygas MH, Brasseaux BK, Moore FA. A multidisciplinary clinical pathway decreases rib fracture-associated infectious morbidity and mortality in high-risk trauma patients. Am J Surg. 2006 Dec;192(6):806-11. doi: 10.1016/j.amjsurg.2006.08.048. PMID 17161098
- [Background] de Jong MB, Kokke MC, Hietbrink F, Leenen LP. Surgical Management of Rib Fractures: Strategies and Literature Review. Scand J Surg. 2014 Jun;103(2):120-125. doi: 10.1177/1457496914531928. Epub 2014 Apr 29. PMID 24782038
- [Background] Shi HH, Esquivel M, Staudenmayer KL, Spain DA. Effects of mechanism of injury and patient age on outcomes in geriatric rib fracture patients. Trauma Surg Acute Care Open. 2017 Mar 16;2(1):e000074. doi: 10.1136/tsaco-2016-000074. eCollection 2017. PMID 29766084
- [Background] Tignanelli CJ, Rix A, Napolitano LM, Hemmila MR, Ma S, Kummerfeld E. Association Between Adherence to Evidence-Based Practices for Treatment of Patients With Traumatic Rib Fractures and Mortality Rates Among US Trauma Centers. JAMA Netw Open. 2020 Mar 2;3(3):e201316. doi: 10.1001/jamanetworkopen.2020.1316. PMID 32215632
- [Background] Pieracci FM, Majercik S, Ali-Osman F, Ang D, Doben A, Edwards JG, French B, Gasparri M, Marasco S, Minshall C, Sarani B, Tisol W, VanBoerum DH, White TW. Consensus statement: Surgical stabilization of rib fractures rib fracture colloquium clinical practice guidelines. Injury. 2017 Feb;48(2):307-321. doi: 10.1016/j.injury.2016.11.026. Epub 2016 Nov 27. No abstract available. PMID 27912931
- [Background] Chen Zhu R, de Roulet A, Ogami T, Khariton K. Rib fixation in geriatric trauma: Mortality benefits for the most vulnerable patients. J Trauma Acute Care Surg. 2020 Jul;89(1):103-110. doi: 10.1097/TA.0000000000002666. PMID 32176172
- [Background] Ryb GE, Dischinger PC, Burch CA, Kerns TJ, Kufera J, Andersen D. Frailty and injury causation. Ann Adv Automot Med. 2012;56:175-81. PMID 23169127
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354
- [Background] Keller BA, Kabagambe SK, Becker JC, Chen YJ, Goodman LF, Clark-Wronski JM, Furukawa K, Stark RA, Rahm AL, Hirose S, Raff GW. Intercostal nerve cryoablation versus thoracic epidural catheters for postoperative analgesia following pectus excavatum repair: Preliminary outcomes in twenty-six cryoablation patients. J Pediatr Surg. 2016 Dec;51(12):2033-2038. doi: 10.1016/j.jpedsurg.2016.09.034. Epub 2016 Sep 28. PMID 27745867
- [Background] Harbaugh CM, Johnson KN, Kein CE, Jarboe MD, Hirschl RB, Geiger JD, Gadepalli SK. Comparing outcomes with thoracic epidural and intercostal nerve cryoablation after Nuss procedure. J Surg Res. 2018 Nov;231:217-223. doi: 10.1016/j.jss.2018.05.048. Epub 2018 Jun 21. PMID 30278932
- [Background] Vossler JD, Zhao FZ. Intercostal nerve cryoablation for control of traumatic rib fracture pain: A case report. Trauma Case Rep. 2019 Jul 31;23:100229. doi: 10.1016/j.tcr.2019.100229. eCollection 2019 Oct. PMID 31388539
- [Background] Koethe Y, Mannes AJ, Wood BJ. Image-guided nerve cryoablation for post-thoracotomy pain syndrome. Cardiovasc Intervent Radiol. 2014 Jun;37(3):843-6. doi: 10.1007/s00270-013-0718-8. Epub 2013 Aug 17. PMID 23954965
- [Background] Byas-Smith MG, Gulati A. Ultrasound-guided intercostal nerve cryoablation. Anesth Analg. 2006 Oct;103(4):1033-5. doi: 10.1213/01.ane.0000237290.68166.c2. PMID 17000825
- [Background] Pieracci FM, Leasia K, Bauman Z, Eriksson EA, Lottenberg L, Majercik S, Powell L, Sarani B, Semon G, Thomas B, Zhao F, Dyke C, Doben AR. A multicenter, prospective, controlled clinical trial of surgical stabilization of rib fractures in patients with severe, nonflail fracture patterns (Chest Wall Injury Society NONFLAIL). J Trauma Acute Care Surg. 2020 Feb;88(2):249-257. doi: 10.1097/TA.0000000000002559. PMID 31804414
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Marasco SF, Martin K, Niggemeyer L, Summerhayes R, Fitzgerald M, Bailey M. Impact of rib fixation on quality of life after major trauma with multiple rib fractures. Injury. 2019 Jan;50(1):119-124. doi: 10.1016/j.injury.2018.11.005. Epub 2018 Nov 3. PMID 30442372
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Derived] Forrester JD, Tung JT, Knight AW, Wang S, Myers AA, King JM, Earley MJ, Guthrie-Baker S, Flojo RB, Chen JT, Abreo AM. Chilling the nerve, easing the pain?: A randomized clinical trial evaluating surgeon-administered bedside percutaneous cryoneurolysis for rib fracture pain. J Trauma Acute Care Surg. 2025 Dec 29. doi: 10.1097/TA.0000000000004885. Online ahead of print. PMID 41604277